CLINICAL TRIAL: NCT00740181
Title: A Phase II Study With Decitabine, Low Dose Cytarabine and G-CSF in High-risk Myelodysplastic Syndromes, Refractory Acute Myeloid Leukemia or Acute Myeloid Leukemia in Patients With Significant Co-morbidities.
Brief Title: Decitabine, Cytarabine, GCSF for Refractory AML/MDS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of efficacy
Sponsor: Brown University (Other)
Collaborators: Memorial Hospital of Rhode Island (Other); Roger Williams Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BrUOG-AML-217; MGI Pharma#DAC 022/2007 (Other: Brown University)
Record Dates: First submitted 2008-08-21; First posted 2008-08-22 (Estimated); Results first posted 2013-07-02 (Estimated); Last update posted 2022-01-14 (Actual); Status verified 2022-01

CONDITIONS: Myelodysplasia; Leukemia
Keywords: myelodysplasia; refractory leukemia; acute leukemia
MeSH Terms: conditions — Anemia, Refractory, with Excess of Blasts; Leukemia | interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Chemotherapy (Experimental): Decitabine 20 mg/m2 IV over 1 hr days 1-5 Cytarabine 20 mg/m2 subcut days 1-5 G-CSF 5mcg/kg subcut days 1-5
  Interventions: Drug: chemotherapy

INTERVENTIONS:
Drug: chemotherapy

SUMMARY:
This study will determine the activity of decitabine, low dose cytarabine (ARA-C) and G-CSF for patients with myelodysplasia and leukemia.

DETAILED DESCRIPTION:
The primary objective of this study is to determine the feasibility and toxicity of decitabine, ARA-C and G-CSF for patients with myelodysplasia, refractory acute leukemia and poor performance status acute leukemia.

ELIGIBILITY:
Inclusion Criteria:

* All patients must have histological confirmation of disease prior to enrollment on study.
* Patients with de novo AML who are not eligible for induction chemotherapy are eligible. Patients with refractory, relapsed AML are eligible.
* Patients with AML evolving from prior MDS or secondary to prior chemotherapy are eligible provided they are not eligible for standard induction chemotherapy.
* Patients with MDS and with blasts > 10% (RAEB-II) are eligible.
* Patients with extramedullary relapse only (i.e., leukemia cutis or other extramedullary site) are eligible as long as disease can be monitored.
* Patients who have relapsed after standard autologous and/or allogeneic bone marrow transplant are eligible as long as they meet all other eligibility criteria.
* Patients must not have had any chemotherapy, except hydrea, or radiation for at least 4 weeks prior.
* Patients must be > 18 years of age.
* Patients with an active second malignancy other than non-melanoma skin cancers are not eligible.
* Patients must have an expected life expectancy of > 12 weeks at the time of enrollment.
* Patients with visceral, blood stream or nervous system opportunistic infection are eligible if the infection has been appropriately treated and controlled. Patients with fungal lung infections must have had treatment for at least one month and have proof of regression prior to enrollment. Patients may be on antimicrobials at the time of therapy.
* Initial required laboratory values:

  * Total Bilirubin < 2 X upper limit of normal.
  * AST & ALT < 3 X upper limit of normal (if elevated liver enzymes thought likely due to Leukemic infiltrate discuss with the Principal Investigator and the BrUOG Central Office).
  * Creatinine < 2 mg/dl.
  * < 15,000 K/uI blast count-Hydroxyurea can be used to decrease count if more than 15,000 K/ul.
* Patients must have an ECOG performance status of 0-2.
* Patients must receive and sign a full informed consent.
* Patients should not have co-existing medical illnesses which would limit survival < 12 weeks.
* No known history of HIV.
* The safety of decitabine in human pregnancy is unknown. Based on animal studies, decitabine may cause fetal harm when administered to a pregnant woman. Therefore, it is important that you do not become pregnant or father a child while receiving study medication and for 2 months afterwards because the drugs in this study may affect an unborn baby.
* If you are a woman capable of becoming pregnant (not surgically sterile or post-menopausal), you must have a negative pregnancy test before beginning treatment.

If you do become pregnant, suspect you are pregnant, or if your partner becomes pregnant while you are on this study, you must notify your study doctor immediately. If you become pregnant, you will be taken off this study.

In addition, you must not breast feed at any time you are on this study since any drugs you are taking may also affect the child.

If you are capable of giving birth to or fathering a child, you must agree to use a form of birth control (examples of effective birth control are: a condom or a diaphragm with spermicidal jelly; oral, injectable, or implanted birth control; or abstinence) that is medically acceptable to your study doctor while taking part in this research study.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2008-08; Primary Completion 2010-02 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Butera, Principal Investigator — Brown University
Locations (1):
- Lifespan Hospitals, Providence, Rhode Island, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 9 patients were enrolled beginning April 2009 to February 2010
Period: Overall Study
Arm/Group | Chemotherapy
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Chemotherapy
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 73 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Response Rate
Description: Complete Response/Complete Remission:
  Complete remission (CR) is defined as the presence of all of the following:
  * Peripheral blood - No leukemic blasts present.
  * No extramedullary findings of leukemia or disappearance of such (i.e. CNS or soft tissue involvement)
  * Bone marrow
  * No Auer rods
  * Less than 5% blast cells.
  * CBC and bone marrow criteria must be met within one week of each other.
  * Hemoglobin 9g/dl or greater
  * Neutrophil count >1000 and platelet count >100,000.
  * RBC Transfusion free for 2 weeks.
Time Frame: within 30 days of last treatment
Measure: Number; unit: participants
Arm/Group | Chemotherapy
Number analyzed (Participants) | 9
participants | 1

ADVERSE EVENTS:
Time Frame: Pre-study and prior to each cycle of treatment (on average for 2 cycles, approximately 8-10 weeks)
Arm/Group | Chemotherapy
Serious Adverse Events (participants affected / at risk) | 8/9
Other Adverse Events (participants affected / at risk) | 0/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chemotherapy (N=9)
fever (Investigations) | 2 (2)
death within 30 days treatment- disease related (Investigations) | 3 (3)
dyspnea/penumonitis and bilateral infiltrates , death within 30 days of treatment (Investigations) | 1 (1) — not related to txt
hemmorrhage-brain, pain-neuro(H/A), weakness (Investigations) | 1 (1)
infection (Investigations) | 1 (1)
acute respiratory failure- death not related, neutropenic fever - not related (Investigations) | 1 (1)
infection, neutropenia (Investigations) | 1 (1)
fever, infection/pulmonary/upper respiratory (pneumonia) (Investigations) | 1 (1)
PLT, hemorrhage bladder & CHF/L ventricular systolic dysfunction, infection-pulmonary (Investigations) | 1 (1) — also: constipation(3), urinary retention(2)
thrombocytopenia, mucositis, dehydration, dysphagia, syncope, anemia (Investigations) | 1 (1)
hypoxic respiratory failure and septic shock- possibly related (Investigations) | 1 (1)
thrombocytopenia, hypoxia, pleural effusion (Investigations) | 1 (1)
syncopal episodes and anemia (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No